CLINICAL TRIAL: NCT00003647
Title: Phase III Randomized Study of Dacarbazine With or Without Allovectin-7 in Patients With Metastatic Melanoma
Brief Title: Chemotherapy With or Without Immunotherapy in Treating Patients With Stage III or Stage IV Melanoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vical (Industry)
Purpose: Treatment
Other Study IDs: CDR0000066736; VCL-1005-301; NCT00416416 (obsolete NCT alias)
Record Dates: First submitted 1999-11-01; First posted 2004-03-23 (Estimated); Last update posted 2008-07-25 (Estimated); Status verified 2008-07

CONDITIONS: Stage IV Melanoma; Stage III Melanoma; Recurrent Melanoma
Keywords: adult solid tumor; body system/site cancer; cancer; melanoma; recurrent melanoma; skin tumor; solid tumor; stage III melanoma; stage IV melanoma; stage, melanoma
MeSH Terms: conditions — Melanoma; Neoplasms; Skin Neoplasms | interventions — Allovectin-7; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: allovectin-7
Drug: allovectin-7/dacarbazine
Drug: dacarbazine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Injecting allovectin-7 into a person's melanoma cells may make the body build an immune response that will kill tumor cells.

PURPOSE: Randomized phase III trial to compare the effectiveness of dacarbazine with or without immunotherapy in treating patients who have stage III or stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Demonstrate either an improvement in the median time to disease progression by at least 2 months with no decrease in the rate of objective clinical response OR an improvement by at least 15% in the rate of objective clinical response with no decrease in the median time to disease progression in patients with stage III or IV melanoma receiving dacarbazine with Allovectin-7 when compared with patients receiving dacarbazine alone.

II. Determine the benefits, risks, and side effects of these regimens in this patient population.

PROTOCOL OUTLINE: This is a randomized, multicenter study. Patients are stratified according to sex, age, and spread of disease (cutaneous or nodal vs visceral disease). Patients are randomized to one of two treatment arms.

Arm I: Patients receive dacarbazine IV over 1 hour on day 0. Arm II: Patients receive treatment as in arm I. Patients also receive Allovectin-7 intratumorally on days 3 and 10.

Patients with stable or responding disease may receive additional courses every 28 days.

Patients are followed every 4 months.

PROJECTED ACCRUAL:

A total of 280 patients (140 in each arm) will be accrued for this study.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Histologically confirmed stage III or IV melanoma 1 or more metastatic tumors for which surgery is not deemed to be a curative option
* Dacarbazine is indicated as first line chemotherapy
* At least 1 measurable tumor at least 1 cm2 but no greater than 100 cm2
* No history of brain metastases

--Prior/Concurrent Therapy--

* Biologic therapy: At least 4 weeks since prior biologic therapy
* Chemotherapy: See Disease Characteristics; No prior chemotherapy
* Endocrine therapy: No concurrent immunosuppressive drugs
* Radiotherapy: At least 4 weeks since prior radiotherapy
* Surgery: At least 2 weeks since prior major surgery
* Other: No other concurrent anticancer drug therapy or experimental therapy

--Patient Characteristics--

* Age: 18 and over
* Performance status: Karnofsky 80-100%
* Life expectancy: At least 24 weeks
* Hematopoietic: WBC at least 3,000/mm3; Platelet count at least 100,000/mm3; Hemoglobin at least 9 g/dL
* Hepatic: Bilirubin no greater than 2.0 mg/dL; SGOT/SGPT less than 3 times upper limit of normal (ULN); PT/PTT normal; Albumin normal; LDH no greater than 2 times ULN
* Renal: Creatinine no greater than 2.0 mg/dL
* Cardiovascular: No uncontrolled hypertension; No New York Heart Association class III or IV disease
* Other: HIV negative; Not pregnant or nursing; Negative pregnancy test; Fertile patients must use effective contraception; No active autoimmune disease; No active infection requiring parenteral antibiotics; No uncontrolled diabetes mellitus; No other prior malignancy within the past 5 years except skin cancer or stage 0-II cervical cancer; No significant psychiatric disorders

Min Age: 18 Years
Age Groups: Adult, Older Adult
Dates: Start 1998-07; Study Completion 2002-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cherie Smith, Study Chair — Vical
Locations (44):
- United States (44):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - Scripps Memorial Hospitals-Stevens Cancer Center - Encinitas, Encinitas, California
  - Kaiser Permanente-Southern California Permanente Medical Group, San Diego, California
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Washington Cancer Institute, Washington D.C., District of Columbia
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Georgia Cancer Specialists, Decatur, Georgia
  - Georgia Cancer Specialists, P.C., East Point, Georgia
  - St. Francis Medical Center, Honolulu, Hawaii
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Lutheran General Hospital, Park Ridge, Illinois
  - Cancer Care Center for Southern Indiana, Bloomington, Indiana
  - Cancer Care Center, New Albany, Indiana
  - Oncology and Hematology Associates, Westwood, Kansas
  - Lucille Parker Markey Cancer Center, University of Kentucky, Lexington, Kentucky
  - Louisiana State University School of Medicine, New Orleans, Louisiana
  - Franklin Square Hospital Center, Baltimore, Maryland
  - Providence Hospital Cancer Center, Southfield, Michigan
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - North Memorial Health Care, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Park Nicollet Clinic, Saint Louis Park, Minnesota
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Billings Interhospital Oncology Project, Billings, Montana
  - Bergan Mercy Medical Center, Omaha, Nebraska
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - HemOnCare, P.C., Brooklyn, New York
  - Arena Oncology Associates, Great Neck, New York
  - Beth Israel Medical Center, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Mid Dakota Clinic, P.C., Bismarck, North Dakota
  - Mid-Ohio Oncology/Hematology, Inc., Columbus, Ohio
  - Toledo Clinic, Inc., Toledo, Ohio
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Danville Hematology and Oncology, Inc., Danville, Virginia
  - Cancer Treatment Centers of America in Hampton Roads, Portsmouth, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin